CLINICAL TRIAL: NCT03226327
Title: A Pilot Trial on Efficacy and Safety of a Formula Salt With Very Low Sodium (Manlikang) in Reducing Salt Intake and Blood Pressure Among Patients With Hypertension in Community
Brief Title: A Pilot Trial of Manlikang in Reducing Salt Intake and Blood Pressure Among Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yangfeng Wu, director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PUCRI20170716
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Hypertension; Hypertension With Abnormal Renal Function
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hypertension patients (Experimental)
  Interventions: Dietary Supplement: formula salt with very low sodium (Brand name: Manlikang)

INTERVENTIONS:
Dietary Supplement: formula salt with very low sodium (Brand name: Manlikang) — hypertension patients will use the formula salt with very low (<20%) sodium （Manlikang) for six weeks, and will be followed up at 1, 2, 4 and 6 weeks to assess the 24-hour urine sodium.

SUMMARY:
This study is a single arm trial with before-after comparison design. Three groups of patients with hypertension will be recruited: not taking antihypertension drugs and having normal renal function, taking antihypertension drugs and having normal renal function, and having abnormal renal function without regards of antihypertension drugs use. Each group includes 30 patients. Based on renal function test, the investigators provide the Manlikang containing potassium chloride to patients with normal renal function, and provide the Manlikang not containing potassium chloride to patients with abnormal renal function. All hypertension patients will use the formula salt with very low sodium (Manlikang) for six weeks, and will be followed up at 1, 2, 4 and 6 weeks. The primary outcome will be the decrease of patients' systolic blood pressure at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 75 years old
* No planning to move out of the community in the next three months
* Not cooking at home less than 3 times or one day during the study
* Willing to participate in the study and sign informed consent

Exclusion Criteria:

* Acute myocardial infarction, history of stroke in the past 3 months, history of malignancy or expected lifetime less than 1 year.
* Hypercortisolism or aldosteronism
* Acute disease, such as upper respiratory infection, fever and diarrhea.
* Incapable of communicating, such as deaf and dumb, dementia, mental disorder.
* Families taking salt substitute currently
* Not willing to use Manlikang in family
* Liver disfunction
* Anyone with abnormal serum potassium in family
* Anyone using potassium-retaining diuretics in family

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
the change of systolic pressure | baseline and 6 weeks
  the change of systolic pressure before and after taking Manlikang

SECONDARY OUTCOMES:
the change in 24-hour urine sodium | baseline and 6 weeks
  the change of 24-hour urine sodium before and after taking Manlikang
incidence of reducing antihypertensive drug dose | up to 6 weeks
  the incidence of reducing antihypertensive drug dose after taking Manlikang in each group.
incidence of reaching the normal blood pressure | up to 6 weeks
  blood pressure reaches the standard of systolic pressure<140mmHg and diastolic pressure<90mmHg after taking Manlikang.
adverse event | up to 6 weeks
  the adverse events after taking Manlikang

CONTACTS AND LOCATIONS:
Locations (1):
- Maoer Shi community, Chongqing, China

REFERENCES:
- [Derived] Liu T, Rao H, Wang M, Xu H, Wang W, Li G, Wang H, Mu L. Comparative analysis of visit and home blood pressure in a pilot trial on the effect of 18% sodium substitute salt on blood pressure. Sci Rep. 2021 Jan 13;11(1):907. doi: 10.1038/s41598-020-79282-2. PMID 33441669
- [Derived] Mu L, Li C, Liu T, Xie W, Li G, Wang M, Wang R, Rao H, He Q, Wang W, Wu Y. A pilot study on efficacy and safety of a new salt substitute with very low sodium among hypertension patients on regular treatment. Medicine (Baltimore). 2020 Feb;99(8):e19263. doi: 10.1097/MD.0000000000019263. PMID 32080135